CLINICAL TRIAL: NCT03479450
Title: Surfactant for Neonatal Respiratory Distress Syndrome at High Altitude Areas:a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Collaborators: the first people hospital of Tibet autonomous region (Unknown); the second people hospital of Lasa (Unknown); the first people hospital of Shigatse (Unknown); the first people hospital of Lasa (Unknown); the people hospital of Linzhi (Unknown); the people hospital of Laqu (Unknown)
Responsible Party: Principal Investigator, Ma Juan, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Other Study IDs: surfactant for NRDS
Record Dates: First submitted 2018-03-18; First posted 2018-03-27 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Surfactant
MeSH Terms: interventions — Surface-Active Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: surfactant — surfactant is given when neonatal respiratory distress syndrome is diagnosed

SUMMARY:
The traditional concept believes that the etiology of neonatal respiratory distress syndrome (RDS) is immature development of lung,especially the surfactant synthesis system,and RDS is still one of the major causes of mortality and morbidity in newborns, especially premature infants.In recent years, using pulmonary surfactant replacement therapy (PS treatment) in the treatment of respiratory distress syndrome (RDS) is a major breakthrough in neonatal medicine.Combined with clinical practice and experience,and through Meta analysis of related randomized controlled trials (RCTs),it confirms that natural surfactant treatment can reduce mortality,the incidence of pulmonary air leaks (pneumothorax and interstitial lung emphysema),and the incidence of bronchopulmonary dysplasia (BPD) or 28-day-old mortality.For RDS in preterm infants whose gestation is <35 weeks ,surfactant replacement therapy is also more effective than in nearly term and full term infants.Therefore, in the analysis of cases of different gestational age groups,the investigators should focus on the study of premature infants cases.Due to less relevant research for using PS treatment to cure newborn RDS in high altitude area,this retrospective study conducts statistics and analysis of recently three-year cases in some hospital of high altitude area,to explore the treatment effect of the high altitude region and the impact of altitude on the treatment.

DETAILED DESCRIPTION:
in order to explore feasibility and efficacy for PS treatment of newborn RDS in high-altitude area ,and its efficacy at different altitudes, the investigators conduct a multi-center retrospective study of RDS cases in Qinghai and Tibet these two high-altitude area,and use RDS cases under the unique conditions to do statistics and analysis.

ELIGIBILITY:
Inclusion Criteria:

* the preterm infants less than 37 weeks were included in the study;diagnosed with NRDS

Exclusion Criteria:

* parents' rejecting to join;major congenital abnormalities

Ages: 10 Minutes to 1 Day | Sex: All
Age Groups: Child
Study Population: the preterm infants less than 37 weeks and diagnosed with NRDS were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
bronchopulmonary dysplasia(BPD) | before discharge or 36 weeks' gestational age
  the incidence of BPD in infants with neonatal neonatal RDS
death | before discharge or 36 weeks' gestational age
  the incidence of BPD in infants with neonatal RDS

SECONDARY OUTCOMES:
intraventriclular hemorrhage(IVH) | before discharge or 36 weeks' gestational age
  the incidence of IVH in infants with neonatal RDS
necrotizing enterocolitis(NEC) | before discharge or 36 weeks' gestational age
  the incidence of NEC in infants with neonatal RDS

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China